CLINICAL TRIAL: NCT00155181
Title: the Garduate Institute of Microbiology in National Taiwan University
Brief Title: Molecular Mechanism of Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Other Study IDs: 9361700387; NHRI-EX94-9419BI
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Epstein-Barr virus; Nasopharyngeal carcinoma; Carcinogenesis
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections; Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
EBV, infection process, immortalization, B lymphocytes, Epithelial cells, co-culture Epstein-Barr virus (EBV) belongs to human γ-herpes viruses. Unlike other human herpes viruses, EBV can only predominately infect two types of human cells: lymphoid cells and epithelial cells and its infection is associated with several human malignancies of these two cell types. The lymphoid cancers associated with EBV infection include Burkitt's lymphoma, Hodgkin's disease, B lymphoma in immunodeficient patients and T/NK cell lymphoma. The carcinomas associated with EBV are nasopharyngeal carcinoma and gastric carcinoma. One unique biological feature of EBV is that it can infect and immortalize primary B lymphocytes in vitro into lymphoblastoid cell lines (LCL). So far, limited information is known about the whole EBV infection process and its regulation mechanism for immortalization. In this project, three EBV infection models are setting up to reveal the cellular events and signal transduction pathway possibly involved in EBV infection process and immortalization course of action.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC), a human malignancy derived from the nasopharyngeal epithelial cells, is occurring highly frequently in Taiwan. Of note, the average ages of NPC individuals are usually ten years younger than those of patients with other head and neck cancers. Clinically, this early onset and high incidence of metastasis in NPC may contribute to its poor prognosis. Fortunately, NPC is usually radio-and chemo-therapy sensitive during the early stage. So, the more we understand NPC pathogenesis, the more efficient detection methods would be developed for NPC early diagnosis and prognosis.

Four unique characteristics have been reported for NPC: geographic preference, heavy infiltration of lymphocytes, high incidence of metastasis and association with Epstein-Barr virus (EBV). According to our hypothesis that both cellular changes and viral factors are crucial for NPC development, four major long-term study goals have been carried out in our lab: (1) identification and characterization of the cellular and viral factors that are involved in NPC formation, (2) elucidation of potencies of these molecules as clinical diagnosis and prognosis markers of NPC, (3) investigation of the molecular and biological linkage between EBV infection and NPC development and (4) establishment of a drug-screening system for NPC chemotherapy.

Based on our assumption that both cellular genes and viral factors are involved in NPC carcinogenesis, the following genes are chosen as the major study targets in this five-year grant. Firstly, to asses the alteration of cellular gene expression, we choose three cytokine genes 【interleukin (IL)-1, IL-7 and IL-13】, three inhibitors of apoptosis proteins (IAP) genes (survivin, HIAP-1, and HIAP-2), two specific cellular genes (osteoblast-specific factor-2 and polymeric immunoglobulin receptor) and one tumor suppressor gene (tumor susceptibility gene TSG101) in our proposal. All these genes exhibit special expression profiles in NPC biopsies in our preliminary study. So, the regulation and effect of these genes in epithelial cells would be the study focus. Secondly, two EBV viral genes, Zta and LMP2A, the former encoded immediately early lytic product and the later encoded latent membrane protein, are selected for this study. In our previous grant, we found that Zta can up-regulate TKT (trk-related tyrosine kinase) and matrix metalloproteinases (MMP)-1 which is a down-stream effector of TKT. Therefore we will extend the study on how Zta and LMP2A regulate and influence anti-apoptotic network and metastasis progression. Based on our preliminary data, this proposal is highly approachable and the results may provide valuable information for NPC diagnosis, prognosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of nasopharyngeal carcinoma

Exclusion Criteria:

-

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hwa Tsai, Ph D, Study Chair — National Taiwan University College of Medicine
Locations (1):
- National Taiwan University College of Medicine, Taipei, Taiwan